CLINICAL TRIAL: NCT04535466
Title: Development of an Artificial Intelligence Precise Diagnosis Predictive Modle for Dense Density Breast Tissue Based on Radiomics
Brief Title: Diagnosis Predictive Modle for Dense Density Breast Tissue Based on Radiomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yaping yang, Clinical Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSU_AI01
Record Dates: First submitted 2020-08-21; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Breast Diseases; Artificial Intelligence; Dense Breast Density; Predictive Cancer Model
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is a prospective, observational cohort study of patients with dense breast tissue. The study was based on the radiomics and other clinicopathological information of patients to establish the diagnostic system for breast disease by using artificial intelligence.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with dense breast density tissue
* Digital breast tomosynthesis was performed
* Breast ultrasound examination was performed
* Pathologic examination of breast lesions was performed

Exclusion Criteria:

* Incomplete clinicopathologic data
* Female patients with fatty glands of the breast

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients aged 18-80 were included in our study who were diagnosed and treated at Sun Yat-sen memorial hospital .
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
the predictive model's area under curve(AUC) | follow up for 2 year for individuals
  To assess the predictive accuracy of the radiomic-based and clinical-based model by using operating characteristic curve (ROC) analysis and calculating the area under the curves (AUC).

CONTACTS AND LOCATIONS:
Locations (1):
- Breast tumor center of Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China